CLINICAL TRIAL: NCT04278794
Title: Optimizing Hospital-to-home Transitions for Older Adults With Stroke and Multimorbidity: A Pragmatic Trial of an Outpatient-based Virtual Transitional Care Intervention
Brief Title: Optimizing Hospital-to-home Transitions for Older Adults With Stroke and Multimorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Hamilton Health Sciences Corporation (Other); Health Quality Ontario (Other); Canadian Frailty Network (Other); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CIHR-419061
Record Dates: First submitted 2020-02-05; First posted 2020-02-20 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Stroke
Keywords: Older adults; Multimorbidity; Transitional care; Virtual care; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Effectiveness-implementation hybrid type I design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Study patients will be blinded to their group allocation. Those aware that they are receiving or not receiving the intervention are more likely to provide biased assessments of the effectiveness of the intervention than blinded participants. Participants who are aware that they are not receiving the intervention may be less likely to comply with the trial protocol, and more likely to drop out of the trial. To minimize assessment bias, Research Assistants will be blinded to group allocation. The statistical analyst will be blinded to the group allocation of the participants when analyzing the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transitional Care Stroke Intervention (TCSI) (Experimental): Participants randomly assigned to the intervention group will be offered the intervention in addition to usual care provided by in-patient and outpatient stroke rehabilitation services. The TCSI is a 6-month stroke transitional care intervention, provided in addition to usual stroke care, that includes four core components: comprehensive hospital discharge plan, structured home visits and telephone support, monthly intraprofessional case conferences, and linkages to primary care and other healthcare and community services. The TCSI will be delivered by an interprofessional team of care providers at the study site, including an occupational therapist, registered nurse, speech language pathologist, physical therapist, and social worker from a hospital-based outpatient stroke rehabilitation setting.
  Interventions: Other: Transitional Care Stroke Intervention (TCSI)
- Control (No Intervention): Usual care provided by in-patient and out-patient stroke rehabilitation services.

INTERVENTIONS:
Other: Transitional Care Stroke Intervention (TCSI) — Core components:
  1. Comprehensive Hospital Discharge Plan. The Care Coordinator will meet with staff in the in-patient unit along with patients and their caregivers to develop and implement a comprehensive discharge plan.
  2. Structured home visits and telephone support. As part of the structured home visits and telephone support, a member of the IP team will provide up to 6 home visits over 6 months. The team will provide: screening and assessment; medication review and reconciliation; self-management support; education; and caregiver assessment.
  3. Monthly IP case conferences. 6 monthly IP team case conferences will be held to discuss goals identified by the patient, collectively develop a plan of care, and identify needs.
  4. Linkages to services. Facilitate timely follow-up with the primary care provider and build relationships with local health and social service providers. These referrals and links will provide the foundation for continued use post-intervention.
  Arms: Transitional Care Stroke Intervention (TCSI)

SUMMARY:
Stroke is the leading cause of death and adult disability in Canada. Sixty percent of these older adults (> 65 years) will return to their homes after a stroke and will require ongoing rehabilitation. About 92% of older adults have two or more chronic conditions. These patients often require services from a number of providers in a number of settings and are therefore, susceptible to fragmented health care when transitioning from hospital to home. New interventions are needed to improve the quality of care as patients move from hospital to home after a stroke. The proposed research project will examine the impact of a new intervention on patient/caregiver health, patient/caregiver and provider experience and costs, compared to usual health care services. The new intervention will be coordinated by a system navigator and consists of four core components: 1) development of a comprehensive discharge plan, 2) up to 6 home visits (supported by phone calls) by an interprofessional outpatient team, 3) monthly case conferences including the interprofessional care team who will discuss and focus on the patient's goals and care needs, and 4) linkages to other healthcare and community services. This multidisciplinary project will build on our previous study, which provided the groundwork for further study of this new intervention.

DETAILED DESCRIPTION:
The overall purpose of this pragmatic randomized controlled trial (RCT) is to adapt, implement and evaluate a novel person- and family-centred Transitional Care Stroke Intervention (TCSI) for older adults (> 55 years) with stroke and multimorbidity (>2 chronic conditions) and their caregivers. The TCSI is a theory- and evidence-based 6-month intervention designed to improve the health, experience, and quality of transitioning from hospital-to-home for this vulnerable population. An effectiveness-implementation hybrid type I design will be used, which will focus primarily on examining the effectiveness of the TCSI on quadruple aim outcomes: (i) patient and caregiver health outcomes, (ii) patient and caregiver experience, (iii) provider/manager experience, and (iv) patient healthcare service use costs, and will also evaluate implementation outcomes (e.g., barriers, facilitators, fidelity). Our earlier pre-post study provided evidence to support the feasibility, acceptability and preliminary effectiveness of the TCSI on reducing hospital readmissions and emergency department visits (for any cause). These improvements were achieved at no additional cost. The key components of the TCSI in this earlier study included home visits supported by telephone calls by an interprofessional team (IP), patient-centered care planning, and care coordination/recruitment. The following enhancements to the TCSI will be included in the trial: 1) integrating the navigator role across the care continuum, 2) testing the TCSI with a larger sample and more rigorous (RCT) design, 3) enhancing patient self-management, and 4) evaluating the impact of the intervention on caregiver health outcomes and experience. These improvements alongside the inclusion of additional evaluation measures will enable rigorous evaluation of the TCSI and position it for future scale-up and spread

ELIGIBILITY:
Inclusion Criteria:

* age 55 years or greater
* hospitalized for stroke and receiving in-patient rehabilitation
* diagnosed with at least 2 or more chronic conditions
* will be discharged to the community from in-patient rehabilitation (not hospital or long-term care)
* not planning to move out of the study catchment area in the next 6 months
* referred to outpatient stroke rehabilitation services
* capable of providing informed consent, or have a substitute decision-maker who is capable and able to provide informed consent on his/her behalf
* competent in English, or has an interpreter who is competent in English

Exclusion Criteria:

* less than 55 years of age
* fewer than two chronic conditions
* planned discharge to hospital or long-term care facility
* cognitively impaired with no substitute decision maker who is capable to provide consent
* not competent in English with no interpreter

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Sex and gender-based analysis will be completed. Particular attention will be given to sex/gender differences in experiences with the care team, given reported differences in how women and men collaborate with healthcare providers. Additionally, sex-based sub-group analysis will be completed because of the central role that sex plays in healthcare research.
Enrollment: 90 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Any hospital readmission for any cause within 6 months | 6-months
  The Health and Social Services Utilization Inventory (HSSUI) will be used to identify patients with any readmission to hospital for any cause within 6 months from study enrolment. The HSSUI is a reliable and valid self-report questionnaire that measures the use of health and social services from a societal perspective. The question in the HSSUI pertaining to any hospital readmission for any cause will be: "Have you been readmitted to the hospital in the past 6-months?" (Yes / No).

SECONDARY OUTCOMES:
Change in health-related quality of life - mental health | Baseline; 6 months
  The Short-Form 12 Health Survey Version 2 (SF-12v2) tool will be used to assess change in mental health. The tool consists of 12 questions that measure functional health and well-being from the participant's perspective. It provides scores for eight health domains (physical functioning, role-physical, bodily pain, general health, social functioning, role-emotional, mental health) by which a psychometrically-based physical component summary and mental component summary score can be calculated. Response options include the frequency of feeling a certain way or behaviour across 3 or 5 categories (e.g., 'all of the time'). Total scale range 0-100. Higher scores represent a better mental health - health-related quality of life. This will be assessed in patients and caregivers.
Change in health-related quality of life - physical health | Baseline; 6 months
  The Short-Form 12 Health Survey Version 2 (SF-12v2) tool will be used to assess change in physical health. The tool consists of 12 questions that measure functional health and well-being from the participant's perspective. It provides scores for eight health domains (physical functioning, role-physical, bodily pain, general health, social functioning, role-emotional, mental health) by which a psychometrically-based physical component summary and mental component summary score can be calculated. Response options include the frequency of feeling a certain way or behaviour across 3 or 5 categories (e.g., 'all of the time'). Total scale range 0-100. Higher scores represent a better physical health - health-related quality of life. This will be assessed in patients and caregivers.
Change in self-efficacy | Baseline; 6 months
  The Stroke Self-Efficacy Questionnaire (SSEQ) will be used to assess change in self-efficacy of the patient. The SSEQ is a 13-item self-report scale measuring self-efficacy judgements in specific domains of functioning post stroke. Individuals rate their belief in their ability to achieve each of the 13 items on a 10-point scale, where 0 = not at all confident to 10 = very confident. A higher score represents a higher self-efficacy. This will be measured in patients.
Change in depressive symptoms | Baseline; 6 months
  The Center for Epidemiologic Studies on Depression 10-Item Scale (CES-D-10) will be used to assess change in depressive symptoms and symptom severity. This tool has been used in prior studies of older adults with mood disorders, has a high degree of reliability and validity, distinguishes between depressed and non-depressed people, and is a sensitive tool for measuring changes in depressive symptoms over time in psychiatric populations. Participants will be asked about the way they have felt or behaved in response to 10 statements such as 'I was happy'. Response options ask participants to select the frequency they have felt or behaved during the last week, ranging from 'rarely or none of the time (less than 1 day)', 'some or a little of the time (1-2 days)', 'occasionally or moderate (3-4 days)', to 'most or all of the time (5-7 days)'. Scale range: 0 - 30. Higher scores represent more depressive symptoms. This will be measured in patients.
Change in anxiety | Baseline; 6 months
  The Generalized Anxiety Disorder 7-Item (GAD-7) will be used to assess change in anxiety symptoms and severity of symptoms. The GAD-7 is a 7-item tool that asks about the type and frequency of being bothered by a list of problems. Response options include 'not at all', 'several days', 'more than half the days', or 'nearly every', over the last two weeks. Scale range: 0 - 21. Higher scores represent more anxiety. This will be measured in patients.
Change in stroke physical function | Baseline; 6 months
  The Stroke Impact Scale (SIS-16) will be used to assess change in physical functional capacity following stroke. The SIS is a self-report questionnaire that evaluates disability and health-related quality of life following stroke. Scores range from 16 to 80, with a higher score indicating a higher level of functional capacity. This will be measured in patients.
Change in community integration | Baseline; 6 months
  The Community Integration Questionnaire (CIQ) will be used to assess change in level of integration in community. The CIQ consists of 15 items relevant to home integration (H), social integration (S), and productive activities (P). Scores range from 0-29 with a higher score indicating a higher level of community integration. This will be measured in patients.
Change in use of health and social services | Baseline; 6 months
  The HSSUI will be used to assess change in use of health and social services of patients and caregivers. The HSSUI is a reliable and valid self-report questionnaire that measures the use of health and social services, from a societal perspective. The HSSUI provides information on different categories of use including acute care service use such as emergency department visits and hospitalizations, use of nursing and allied health professionals, and visits to family doctors and specialists. Change in the use of health and social services will be assessed for patients and caregivers using the HSSUI.
Change in caregiver strain | Baseline; 6 months
  The Modified Caregiver Strain Index (MCSI) will be used to assess change in caregiver strain. This tool will ask caregivers a list of 13 activities that they may have found to be difficult such as sleeping, physical strain, financial strain, personal plans, and work and family adjustments as a result of the caregiver role. Response options include 'yes' according to two levels, either 'yes, on a regular basis' or 'yes, sometimes', or alternatively, 'no'. Scale range: 0 - 26. Higher scores represent more strain. This will be assessed in caregivers.
Relative risk of any hospital readmission for any cause within 6 months | Baseline; 6 months
  The Health and Social Services Utilization Inventory (HSSUI) will be used to assess any readmission to hospital for any cause (patient). The HSSUI is a reliable and valid self-report questionnaire that measures the use of health and social services from a societal perspective. The HSSUI provides information on different categories of use including acute care service use such as emergency department visits and hospitalizations, use of nursing and allied health professionals, and visits to family doctors and specialists. The relative risk of any hospitalization within six months for any cause will be examined for patients in the intervention group compared to patients in the control group.
Time to any hospital readmission for any cause within 6 months | Baseline; 6 months
  Data from the Institute for Clinical and Evaluative Sciences (IC/ES) will be used to assess the time to any hospital readmission for any cause for patients. The Hospital Discharge Abstract Database (DAD) within IC/ES will be used to measure readmission.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Markle-Reid, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - Hotel Dieu Shaver, Saint Catherines, Ontario

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

REFERENCES:
- [Derived] Markle-Reid M, Fisher K, Walker KM, Beauchamp M, Cameron JI, Dayler D, Fleck R, Gafni A, Ganann R, Hajas K, Koetsier B, Mahony R, Pollard C, Prescott J, Rooke T, Whitmore C. The stroke transitional care intervention for older adults with stroke and multimorbidity: a multisite pragmatic randomized controlled trial. BMC Geriatr. 2023 Oct 24;23(1):687. doi: 10.1186/s12877-023-04403-1. PMID 37872479